CLINICAL TRIAL: NCT07182045
Title: Impact of Uterine and Ovarian Vessel Occlusion on Blood Loss in High Burden Minimally Invasive Myomectomy.
Acronym: Myo-Bleed
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Randa Jalloul, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-25-0413
Record Dates: First submitted 2025-09-16; First posted 2025-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Myoma; Surgery
Keywords: myoma; blood loss
MeSH Terms: conditions — Myoma; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temporary vessel clamps (Experimental): Use of temporary laparoscopic vessel clamps on uterine and ovarian vessels
  Interventions: Other: Temporary clamping of uterine and ovarian vessels
- No Temporary vessel clamps (No Intervention): No use of vessel clamps

INTERVENTIONS:
Other: Temporary clamping of uterine and ovarian vessels — Surgeon will temporarily clamp uterine and ovarian vessels.
  Other Names: Vessel occlusion
  Arms: Temporary vessel clamps

SUMMARY:
This study hypothesizes that temporary bilateral uterine and utero-ovarian artery occlusion with laparoscopic clamps at time of minimally invasive myomectomy will lead to a decreased blood loss at time of myomectomy compared to minimally invasive myomectomy without temporary occlusion.

DETAILED DESCRIPTION:
Background: Leiomyomas are the most common benign tumor of the uterus and affect approximately 70-80% of the population with a uterus . Patients who opt to undergo treatment for a fibroid uterus have a variety of options including medical management, embolization, or surgical management; Historically surgical management involved hysterectomy; however, myomectomy has become more popular as a uterine sparing option. Current data supports that minimally invasive myomectomy is associated with lower morbidity and blood loss than traditional abdominal surgery. With advances in Minimally invasive myomectomy (MIS). There continues to be interest in methods to better improve intraoperative and postoperative outcomes. There is currently support for universal use of intramural vasopressin at time of myomectomy and a growing body of evidence to support temporary bilateral occlusion of the uterine and/or uteroovarian arteries at time of myomectomy to decrease blood loss.

High myoma burden is associated with an increased blood loss at time of surgical management.

Previous studies assessing the utility in temporary occlusion of the uterine and/or utero-ovarian vessels have not specifically evaluated the impact on high myoma burden individuals. As higher myoma burden is addressed in a minimally invasive fashion, it is important to specifically evaluate techniques to optimize these procedures. This study will specifically evaluate the effect of temporary bilateral uterine artery and utero-ovarian occlusion with laparoscopic clamps at the time of minimally invasive myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing minimally invasive myomectomy with either a single intramural or Submucosal fibroid =/>5cm or
* Patients undergoing minimally invasive Myomectomy with =/> 5 fibroids

Exclusion Criteria:

* Pregnancy,
* Age <18yo,
* Patients undergoing concomitant surgery such as endometriosis surgery,
* Suspected malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with female reproductive organs
Enrollment: 120 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Estimated blood loss | Intraoperative (during surgery, which is < 24 hours)
  Estimated blood loss during the surgery between groups, calculated by suction prior to irrigation.

IPD SHARING:
Plan to Share IPD: No